CLINICAL TRIAL: NCT05186142
Title: Interest of the Ultrasound Follow-up of Lymphedema by Elastography Assessment and Cutaneous and Subcutaneous Thickness Measurement During Intensive Treatment of Lymphedema.
Brief Title: Tissue Elastography Assessement and Cuteous and Cubcutaneous Thickness Measurement Following Manual Lymph Drainage in Legs With Lymphedema
Acronym: ELASTOLYMPH
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL19_0482
Record Dates: First submitted 2021-11-12; First posted 2022-01-11 (Actual); Last update posted 2022-01-11 (Actual); Status verified 2021-12

CONDITIONS: Lymphedema; Lower Limb Lymphedema
Keywords: Skin suppleness; Elastography; lymphedema; Manual Lymphatic Drainage
MeSH Terms: conditions — Lymphedema | interventions — High-Energy Shock Waves

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients hospitalized for treatment of lymphoedema: Patients hospitalized for treatment of lymphoedema
  Interventions: Other: Ultrasonography / Ultrasound elastography

INTERVENTIONS:
Other: Ultrasonography / Ultrasound elastography — Ultrasonography / Ultrasound elastography

SUMMARY:
Tissue Elastography Assessement and Cuteous and Cubcutaneous Thickness Measurement Following Manual Lymph Drainage in Legs With Lymphedema

Hence the importance of evaluating the impact of an intensive five-day decongestive treatment on lymphedema in terms of cutaneous flexibility and edema regression.

Patients who are undergoing intensive decongestive treatment for four or five days in the department perform an ultrasound check/examiantion on the first day.

During this echography, in 5 usual measurement points are made an ultrasound image recording (for measurement of cutaneous and subcutaneous thicknesses) and an elastography sequence (an instantaneous measurement).

The study hypothesis is to note that intensive decongestive treatment has an impact on tissues flexibility and cutaneous and subcutaneous thickness.

No many authors discussed this suject, hence the interest of this study. All the data collected and the results obtained will serve for further studies.

ELIGIBILITY:
Inclusion criteria:

* Major patients with unilateral or bilateral lymphedema of the lower limb (s), stage II or III, of primary or secondary origin
* Major patients with admitted for the realization of an Intensive Decongestive Treatment (TDI) of three to five days in the lymphology unit of the Saint Eloi hospital, of Montpellier UHC.

Exclusion criteria:

* Patients with different lymphedema localisation than the lower limbs
* Patient with amputated
* patient not consenting or included in another clinical research study.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients receinving intensive treatment for lower limb lymphedema at UHC Saint Eloi.
  Patients with lower limb lymphedema coming to UHC Saint Eloi for intensive treatment.
Sampling Method: Non-Probability Sample
Enrollment: 47 (Actual)
Dates: Start 2019-05-01 (Actual); Primary Completion 2019-08-01 (Actual); Study Completion 2019-10-20 (Actual)

PRIMARY OUTCOMES:
number of Elastography | day 1 (pre treatment)
  number of Elastography
number of Elastography | day 5 (post treatment)
  number of Elastography

SECONDARY OUTCOMES:
number of Cutaneous thicknesses | day 1 (pre treatment)
  number of Cutaneous thicknesses
number of Cutaneous thicknesses | day 5 (post treatment)
  number of Cutaneous thicknesses
number of Subcutaneous thicknesses | day 1 (pre treatment)
  number of Subcutaneous thicknesses
number of Subcutaneous thicknesses | day 5 (post treatment)
  number of Subcutaneous thicknesses
number of Limb volumetry | day 1 (pre treatment)
  number of Limb volumetry in milliliter
number of Limb volumetry | day 5 (post treatment)]
  number of Limb volumetry in milliliter

CONTACTS AND LOCATIONS:
Overall Officials: MESTRE GODIN Sandrine, Study Director — University Hospital, Montpellier
Locations (1):
- Uhmontpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC